CLINICAL TRIAL: NCT04213053
Title: Changes in Range of Ocular Motility Following Horizontal Rectus Muscle Surgery in Concomitant Strabismus; a Quantitate Measurements Using Lees Screen
Brief Title: Lees Screen in Concomitant Strabismus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farag Khalil Ibrahiem, Assistant Professor, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Paediatric ophthalmology unit
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Intervention Model Description: detect if there are any change in motility after concomitant horizontal muscle surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concomitant strabismus patients (Other): Horizontal strabismus surgery
  Interventions: Procedure: strabismus surgery

INTERVENTIONS:
Procedure: strabismus surgery — Lees screen before and after concomitant strabismus surgery

SUMMARY:
Preoperative and postoperative Lees screen was done after concomitant horizontal strabismus surgery to detect any limitation in the field of operated muscle

DETAILED DESCRIPTION:
Preoperative and postoperative Lees screen was done for concomitant esotropia and exotropia patients to record any change in ocular motility as regards underaction or overaction in the operated extra ocular muscles

ELIGIBILITY:
Inclusion Criteria:

* Concomitant esotropia
* Concomitant exotropia
* Above 10 years old patients

Exclusion Criteria:

* Restrictive and paralytic strabismus
* Previous strabismus surgery
* Mental disability

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
postoperative Lees screen | 3 months
  detect any restriction in muscle field

CONTACTS AND LOCATIONS:
Overall Officials: Sahar TA Abdelaziz, MD, Principal Investigator — Minia University
Locations (1):
- Faculty of Medicine, Minya, Minya Governorate, Egypt